CLINICAL TRIAL: NCT06156293
Title: Prevention of Insomnia Using a Stepped Care Model in Adults: a Pragmatic Stepped-wedge Cluster Randomized Trial
Brief Title: Prevention of Insomnia Using a Stepped Care Model in Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CHAN NGAN YIN, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20230816.02
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disturbance
Keywords: Sleep Disturbance; Stepped care model; Stepped wedge cluster randomized trial; Prevention program
MeSH Terms: conditions — Parasomnias | interventions — Annexin A5

STUDY DESIGN:
Intervention Model Description: Pragmatic stepped wedge design - over 4 months, 18 sites enter trial at 1 month intervals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stepped-care CBT-I group (Experimental): A total of 3 steps of sleep focused intervention will be provided, with the objectives to increase the awareness of sleep health, increase sleep literacy, establish good sleep hygiene and treat insomnia.
  Step 1: self-help digital sleep focused program; Step 2: guided intervention; Step 3: individualized consultation.
  Interventions: Behavioral: Cognitive behavioral prevention program for insomnia (CBP-I)
- Control group (No Intervention): Participants in the control group remain unexposed to the stepped-care sleep-focused intervention.

INTERVENTIONS:
Behavioral: Cognitive behavioral prevention program for insomnia (CBP-I) — CBP-I will be provided to participants once their districts are exposed.
  Arms: Stepped-care CBT-I group

SUMMARY:
Insomnia is one of the most common sleep disorders and affects approximately 10 - 40% of the population across different age groups in Hong Kong. Our previous study has shown that insomnia can be prevented through a brief cognitive behavioral prevention program in adolescents. However, there is very limited data in the adult population.

Current study aims to evaluate a digital sleep-focused platform which consists of different intervention plan according to user's insomnia severity level and employed a stepped care model. Thus, the effectiveness of the stepped care model will be evaluated in a real world setting using stepped wedge cluster randomized controlled design to evaluate potential preventive effect on adults who only with mild insomnia symptoms. The program will be rolled out to different districts in Hong Kong sequentially in 18 districts over 4 steps with a equally spaced time periods. The primary aim of this study is to evaluate the effects of a stepped-care CBT-I model in improving sleep and prevent the incidence of insomnia among participants with mild insomnia.

DETAILED DESCRIPTION:
This interventional study will be a multicenter, assessor-blinded, pragmatic stepped-wedge cluster randomized controlled trial. A total of 18 districts will be included in the study and the randomization will be carried out based on the districts. The stepped-care CBT-I intervention will be sequentially rolled out to the 4-6 districts per step according to a computer-generated random number while the remaining clusters will continue to stay unexposed to the CBT-I intervention over the control period. Therefore after 4-step exposure, all clusters will receive the stepped-care CBT-I intervention. A total of 3 follow-up assessments (post intervention, 3-month and 12-month follow up) will be conducted to assess the effectiveness and long-term effects of the stepped care model.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese adults aged 18-70 years old,
2. The score of Insomnia Severity Index < 10.

Exclusion Criteria:

1. present with psychotic disorders such as bipolar disorder and schizophrenia,
2. present with severe depression or suicidal ideation,
3. present with neurodegenerative diseases that prevent participant from completing the intervention (e.g., dementia and Parkinson's disease).
4. unable to provide consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1016 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Insomnia severity index | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month postintervention and 12-month post-intervention follow up
  The primary outcome will be the perceived insomnia severity measured by Insomnia Severity Index (ISI).

SECONDARY OUTCOMES:
Severity of depression | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  Patient Health Questionnaire-9 (PHQ-9) will be used to measure the severity of depression.
Severity of anxiety | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  General Anxiety Disorder-7 (GAD-7) will be used to measure the severity of anxiety.
Health-related quality of life | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  The health-related quality of life (HRQoL) will be measured by the EuroQol-5D (EQ).
Chronic insomnia diagnosis | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  A checklist based on Diagnostic and statistical manual of mental disorders will be implemented to measure the incidence of chronic insomnia.
Medication usage | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  A checklist will be used to measure the subject's medication usage change.
Clinical global impression | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  Clinical Global Impression (CGI) will be used to assess the insomnia severity over time.
Patient-report clinical global impression | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  A single-item CGI will be used to ask the participant whether they experience sleep improvement or change over the past week or not.
Sleep duration | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  Two self-report questions will be used to record the sleep duration during weekdays and weekends of the participants.
Subjective sleep as measured by sleep diary | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  Self-report sleep diary will be used to record subjective sleep of the participants including total time in bed, sleep onset latency, total sleep duration, sleep efficiency and wake after sleep onset.
Healthcare resource use | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  The use and expense of sleep-promoting medication, psychotherapy, and other complementary treatments for sleep improvement will be collected from individual participants using a self-developed questionnaire, with a focus on their healthcare resource utilization.
Work and social functioning | Post-intervention (ranging from 8 weeks to 24 weeks, depending on the treatment level), 3-month post-intervention and 12-month post-intervention follow up
  A 5-item questionnaire developed from Work and Social Adjustment Scale (WSAS) will be used to measure the daytime functioning of the participants such as ability to work, home management, social and private leisure activities, and close relationship maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Yun Kwok Wing, FRCPsych, Principal Investigator — Department of Psychiatry, the Chinese University of Hong Kong
Locations (1):
- Department of Psychiatry, the Chinese University of Hong Kong, Hong Kong, China